CLINICAL TRIAL: NCT03239418
Title: A Novel Treatment Using Neuromuscular Electrical Stimulation to Improve Eyelid Function in Patients With CN III and CN VII Palsy.
Brief Title: NMES to Improve Eyelid Functions in Cranial Nerve (CN) III and VII Palsy
Acronym: EyeStim
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRCRC2016_001
Record Dates: First submitted 2017-07-31; First posted 2017-08-04 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Blepharoptosis; Lagophthalmos
Keywords: NMES
MeSH Terms: conditions — Blepharoptosis; Lagophthalmos

STUDY DESIGN:
Intervention Model Description: Active treatment vs. Sham control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants in treatment and sham group undergo all of the same procedures except a sham NMES treatment is provided to the control group. Only the treating clinician is aware of group allocation. The investigator and outcomes assessor are unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EyeStim Group (Experimental): Receive an active NMES treatment to the targeted muscles controlling eyelid function.
  Interventions: Device: Neuromuscular electrical stimulation
- Control Group (Sham Comparator): Undergo all the same procedures as the EyeStim group except receive a sham NMES treatment.
  Interventions: Device: Sham neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — A low level electrical current is applied to the muscle that control eyelid function through small electrodes applied to the skin over the target muscles. Treatment is applied daily for 5 consecutive days and exercises for eyelid function are performed in conjunction with the stimulation.
  Arms: EyeStim Group
Device: Sham neuromuscular electrical stimulation — Electrodes are applied to the skin over the target muscles and patient perform the exercises for eyelid function for 5 consecutive days just as in the experimental group, However participants do not receive the electrical stimulation. Due to the low intensity of the stimulation all participants regardless of group allocation are told they may or may not feel the electrical stimulation.
  Arms: Control Group

SUMMARY:
Traumatic brain injury, stroke and other neurological conditions may result in weakness of the muscles that either open or close the eye. This is generally a result of impaired functioning of the oculomotor or facial cranial nerves. Current treatments to improve eye opening or closing are either invasive or largely ineffective. This study tests a noninvasive means of improving eyelid opening and closing by applying a previously demonstrated safe and effective neuromuscular electrical stimulation (NMES) intervention to the muscles controlling eyelid movement. Participants in this study will either receive the investigational NMES protocol 30 min per day for five days or a sham NMES for the same period. The primary outcome for this study is the participants' ability to open or close their affected eye. Secondary outcomes include additional measures of eye and corneal health.

ELIGIBILITY:
Inclusion Criteria:

* Cranial nerve III (oculomotor nerve) and/or cranial nerve IV (facial nerve) palsy.
* Able to read and communicate in English.

Exclusion Criteria:

* Idiopathic onset of CN III and/or CN IV palsy.
* Traumatic injury to the eye or eyelid.
* Active wounds in the treatment area.
* Presence of swelling or infection in or surrounding the affected eye.
* Diminished sensation in the area to be treated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Marginal reflex distance-1 (MRD-1) | Within 1 week of last treatment session.
  Measure of eyelid function for participants with CN III or CN VII palsy
Palpebral fissure height | Within 1 week of last treatment session.
  Measure of eyelid function for participants with CN III or CN VII palsy

SECONDARY OUTCOMES:
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Within 1 week of last treatment session.
  Measure of Quality of Life for participants with CN III or CN VII palsy
Upper eyelid crease distance | Within 1 week of last treatment session.
  Measure of eyelid function in participants with CN III or CN VII palsy

OTHER OUTCOMES:
Distance visual acuity | Within 1 week of last treatment session.
  Measure of overall eye health and function
Distance alternate cover test. | Within 1 week of last treatment.
  Measure of overall eye health and function
Pupil test | Within 1 week of last treatment session.
  Measure of overall eye health and function
Oculomotor exam | Within 1 week of last treatment session.
  Measure of overall eye health and function in participants with CN III palsy
Cornea, Static Asymmetry, Dynamic Function, Synkinesis Classification Scale (CADS). | Within 1 week of last treatment session.
  Measure of ophthalmic involvement in facial function in participants with CN VII palsy

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ngo, MD, Principal Investigator — Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No